CLINICAL TRIAL: NCT03302429
Title: Evaluation of Platelet-rich Fibrin / Biphasic Calcium Phosphate Effect Versus Autogenous Bone Graft on Reconstruction of Alveolar Cleft Defect in the Maxillary Arch: Randomized Controlled Clinical Trial
Brief Title: Evaluation of Platelet Rich Fibrin / Biphasic Calcium Phosphate Effect Versus Autogenous Bone Graft on Reconstruction of Alveolar Cleft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebatallah G Samra El-Shamy, resarcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-09-31
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2017-10

CONDITIONS: Alveolar Ridge Abnormality
Keywords: Alveolar cleft -Platelet rich fibrin- calcium phosphate
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Eighteen patients will be divided into two equal groups. Each group comprises nine patients.
  Group A: Platelet-rich Fibrin combined with Biphasic Calcium Phosphate.(interventional group) Group B: autogenous bone graft (controlled group)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF/ BCP (Experimental): Biphasic calcium phosphate (BCP)"bioceramic bone substitute combined with platelet rich fibrin PRF
  Interventions: Other: PRF/ BCP
- autogenous bone graft (Active Comparator): Autogenous bone graft involving utilizing bone obtained from the same individual receiving the graft
  Interventions: Other: Autogenous bone graft

INTERVENTIONS:
Other: PRF/ BCP — Platelet rich fibrin combined with biphasic calcium phosphate(experimental group)
  Other Names: Easy-graft/BCP
  Arms: PRF/ BCP
Other: Autogenous bone graft — Bone obtained from the same individual who receiving the graft
  Arms: autogenous bone graft

SUMMARY:
P- Maxillary alveolar cleft defects I- Platelet-rich fibrin (PRF) combined with biphasic calcium phosphate (BCP) C- Autogenous bone graft O- Outcome measure : bone height, bone volume, hospital stay, operation duration T- 6 months S- Randomized controlled clinical trial this study aimed to answer a clinical question whether the use of Platelet-rich Fibrin (PRF) combined with Biphasic Calcium Phosphate (BCP), can be an alternative to autogenous bone graft in reconstruction of alveolar cleft defect in maxillary arch.

DETAILED DESCRIPTION:
this study aimed to answer a clinical question whether the use of Platelet-rich Fibrin (PRF) combined with Biphasic Calcium Phosphate (BCP), can be an alternative to autogenous bone graft in reconstruction of alveolar cleft defect in maxillary arch

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from maxillary alveolar cleft
* Patients' age 8 years and older

Exclusion Criteria:

* Syndromic cases will be excluded
* Patients suffering from platelets disorders.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-19 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
bone height | six months postoperative.
  the vertical bone height measured from the most coronal level of the pyriform aperture to the most apical level of the bony bridge.

SECONDARY OUTCOMES:
bone volume | six months postoperative.
  V= (A1xT) + ( A2 xT) + …….+ (An xT) where:
  V= volume A= area T= thickness of the axial C.T slice N=number of slices
operation duration | within 4 hours ( the actual number of hours will be determined intra-operative )
  It is the time elapsed between using the scalable for incision and the last stitch.
  It will be measured by watch in hours.
hospital stay | within 7 days
  Number of days that patients spend in hospital. Measured by calendar, starting from time of admission ending with time of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt